CLINICAL TRIAL: NCT01190982
Title: A Multicenter, Open-Label, Phase II Study of LEP-ETU for Efficacy and Safety in Patients With Metastatic Breast Cancer
Brief Title: Efficacy and Safety Study of LEP-ETU to Treat Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEP-ETU 202
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LEP-ETU (Experimental): All patient will have baseline to confirm disease status. The disease progression/response is assessed inaccordance to the RECIST guidelines
  Interventions: Drug: LEP-ETU

INTERVENTIONS:
Drug: LEP-ETU — 275 mg/m2, IV (in the vein) on day 1 of each 21 day cycle, 6 Cycles or until progression or unacceptable toxicity develops.
  Other Names: Liposome Entrapped Paclitaxel Easy to Use

SUMMARY:
LEP-ETU is a novel, proprietary delivery system of paclitaxel developed by NeoPharm, Inc. Paclitaxel (currently marketed as Taxol) is an anti-microtubular network agent and is active in a broad spectrum of malignancies. Paclitaxel has poor solubility. In order to enhance the solubility, this drug is formulated with polyoxyethylated castor oil, which leading to infusion-related hypersensitivity reactions. The NeoPharm LEP-ETU is formulated with a mixture of well characterized, synthetic phospholipids and cholesterol. This design eliminates the need for the oil. The LEP-ETU formulation has improved safety profile that is necessary for administering higher doses than would commonly be used with Taxol. The clinical evidence obtained from the NeoPharm Phase I study shows LEP-ETU is better tolerated than Taxol, as indicated by a higher maximum-tolerated dose (MTD). The current Phase II study is designed to accomplish the following objectives:

1. Assess the Overall Response Rate (ORR) of patients with metastatic breast cancer after administered over 90 minutes at the dose of 275 mg/m2 LEP-ETU
2. To evaluate the Progression-Free Survival (PFS)
3. To evaluate the safety of LEP-ETU at 275 mg/m2 level, in particular peripheral neuropathy
4. To evaluate the Overall Survival (OS)

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older and female.
2. Have histologically or cytologically confirmed diagnosis of invasive adenocarcinoma originating in the breast.
3. Have at least one target lesion per RECIST criteria
4. If the patient has received adjuvant or neoadjuvant taxane therapy, the patient must not have relapsed with breast cancer within one year of completing this therapy.
5. Have received prior chemotherapy in the adjuvant or metastatic setting with an anthracycline unless contraindicated.
6. Have no other malignancy within the past five years, except non-melanoma skin cancer, cervical intraepithelial neoplasia (CIN), or in-situ cervical cancer (CIS).
7. Have the following hematology levels at Baseline:

   * ANC greater than or equal to 1,500 x 106 cells/L;
   * Platelets greater than or equal to 100 x 109 cells/L;
   * Hgb greater than or equal to 90 g/L.
8. Have the following chemistry levels at Baseline:

   * AST (SGOT), ALT (SGPT) less than or equal to 2.5 x ULN if no evidence of liver metastases;
   * AST (SGOT), ALT (SGPT) less than or equal to 5 x ULN if liver metastases are present;
   * Total bilirubin less than or equal to 26 micromol/L (1.5 mg/dL);
   * Creatinine less than or equal to 177 micromol/L (2 mg/dL); or 24-hour
   * Alkaline phosphatase less than or equal to 5 x ULN (unless bone metastasis is present in the absence of liver metastasis).
9. Have a life expectancy of greater than or equal to 12 weeks.
10. Have an ECOG Performance status of 0-2.
11. Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment.
12. Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee -approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

1. Patient has radiographic evidence of active (symptomatic, untreated) intraparenchymal brain metastases; any leptomeningeal metastases; or asymptomatic untreated intraparenchymal brain metastases requiring treatment.
2. Patient has received more than 1 prior treatment with a non-taxane agent in the metastatic setting.
3. The only evidence of metastasis is lytic or blastic bone metastases or pleural effusion or ascites.
4. Patient has a known infection with human immunodeficiency virus or active viral hepatitis.
5. Patient has active heart disease including myocardial infarction or congestive heart failure within the previous 6 months, symptomatic coronary artery disease, or uncontrolled arrhythmias.
6. Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug (e.g., uncontrolled bleeding or bleeding diathesis).
7. Any active infection requiring parenteral or oral antibiotics.
8. The patient receives treatment with any:

   * Hormonal or other non-investigational agent therapy within 2 weeks prior to first dose of study drug;
   * Herceptin, mitomycin, or nitrosoureas therapy within 6 weeks prior to first dose;
   * Chemotherapy (except for palliative bisphosphonate therapy for bone pain which can be administered as clinically indicated) within 4 weeks prior to first dose study drug;
   * Investigational drug or immunotherapy within 4 weeks prior to first dose study drug;
   * Concurrent radiation therapy (except for palliative radiotherapy for
   * Radiation therapy within 4 weeks prior to first dose of study drug.
9. Patient has pre-existing peripheral neuropathy of NCI-CTCAE Grade >1.
10. Patient has received paclitaxel, docetaxel, or Abraxane because of metastatic carcinoma.
11. Known hypersensitivity to paclitaxel, Cremophor EL, or liposomes.
12. Pregnant or nursing female patients.
13. Unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assessment of Overall Response Rate (ORR) following treatment of LEP-ETU at 275 mg/m2 dose | 2 years
  The time frame is average. The patient will be treated once every 21 day cycle for 6 cycles. Disease status and tumor response/progression will be assessed based on the Response Evaluation Criteria in Solid Tumor (RECIST) after 2, 4 and 6 cycle. Patient will be followed for overall survival until death.

SECONDARY OUTCOMES:
LEP-ETU 275mg/m2 Induce Progression-Free Survival Assessment | 2 years
  The time frame is average. The patient will be treated once every 21 day cycle for 6 cycles. Disease progression will be assessed after 2, 4 and 6 cycle. Patient will be followed for overall Survival until death.

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Indo-American Cancer Institute and Research Center, Banjara Hills, Hyderabad
  - P.D. Hinduja Antional Hospital & Medical Research Center, Mahīm, Mumbia
  - Jaslok Hospital and Research Center, Mumbai